CLINICAL TRIAL: NCT03167268
Title: Double-blind, Phase II Study to Assess the Effectiveness of Lycopene vs Placebo to Reduce Skin Toxicity in Patients With Colorectal Carcinoma Treated With Panitumumab
Brief Title: Panitumumab Skin Toxicity Prevention Trial
Acronym: PaSTo
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ospedale San Carlo Borromeo (Other)
Responsible Party: Principal Investigator, DR. MAURO MORONI, Director of Oncology Unit, Ospedale San Carlo Borromeo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PaSTo
Record Dates: First submitted 2017-02-27; First posted 2017-05-25 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Colorectal Cancer Metastatic; Skin Toxicity
Keywords: Lycopene; Anti EGFR therapy
MeSH Terms: interventions — Lycopene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lycopene 20mg cpr/die (Experimental): Lycopene is a compound belonging to carotenoid group, largely contained in tomatoes and their derivatives, which has an extreme antioxidant activity. In Dermatology, prolonged use of β-carotenoids in general and of lycopene in particular in the diet showed to be effective in skin protection from ageing, sunlight and radiotherapy damages because these compounds may accumulate in skin and thus contribute to reduce free radicals and inflammation effects.
  Interventions: Drug: Lycopene
- Placebo (Placebo Comparator): Containing same excipients than the experimental "Lycopene 20 mg" but not active principle (Lycopene)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lycopene
  Arms: Lycopene 20mg cpr/die
Other: Placebo
  Arms: Placebo

SUMMARY:
Background and rationale: EGFR represents the main and more studied signal activation pathway in the development of colorectal carcinoma. KRAS, NRAS, BRAF and PI3KA mutations and ERBB2 and MET amplification are responsible for most of the cases of primary resistance to anti-EGFR antibody treatments. Despite the identification of these resistance mechanisms, a primary resistance to the therapy was detected in a certain percentage of cases, in which tumour bio-molecular characteristics would suggest a possible response to anti-EGFR antibody treatment. In these cases, pathway activation mechanisms should exist, which act in an alternative, complementary or parallel way than the EGFR one, allowing tumour progression despite of EGFR pharmacological deactivation. Skin toxicity is a characteristic of drugs having EGFR as a target and it shows itself mainly as a sterile acneiform folliculitis together with neutrophils perifollicular infiltrates but also as skin xerosis and paronychia starting from the earliest cycles of treatment. This skin toxicity seems to be closely related to EGFR activation of pro-inflammatory cytokines able to activate specific inflammatory activators, which induce neutrophils granulocytes chemotaxis. Lycopene is a compound belonging to carotenoid group, largely contained in tomatoes and their derivatives, which has an extreme antioxidant activity. In Dermatology, prolonged use of β-carotenoids in general and of lycopene in particular in the diet showed to be effective in skin protection from ageing, sunlight and radiotherapy damages because these compounds may accumulate in skin and thus contribute to reduce free radicals and inflammation effects. Moreover, lycopene ability to induce apoptosis and to inhibit cell cycle progression in some types of tumour cells, both in vitro and in vivo, has already been described. Lycopene seems to be able to suppress significantly PCNA (Proliferating cell nuclear antigen, cofactor of DNA polymerase-β) and β-catenin nuclear expression in neoplastic cells, essential substrate of WNT/β-catenin pathway, which is itself closely connected to activating pathways often involved in carcinogenesis of some kinds of tumours, in particular of colorectal carcinoma, like Akt/GSK3β/β-catenin and Hippo pathways. For its proved skin anti-inflammatory activity as powerful free radicals scavenger, lycopene, which accumulates itself specifically in skin, could be effective in reducing anti-EGFR drugs toxicity. Contemporary use of lycopene could have a positive effect on anti-EGFR drugs treatment effectiveness in patients with metastatic colorectal carcinoma due to its ability to interfere with pathways involved in neoplastic cells proliferation.

Estimated population:100 patients (50 for each of the two groups of treatment)

Study Framework: In this study, patients suffering from metastatic colorectal cancer and submitted to therapy with panitumumab would be enrolled. According to indications, panitumumab would be used:

in first line combined with Folfox or Folfiri;

in second line combined with Folfiri or treatments containing Irinotecan

in monotherapy in any therapeutic line in patients resistant to Fluoropyrimidines, Oxaliplatin and Irinotecan or intolerant to these drugs.

Standard schedules of these treatments would be used.

This is a phase-II, randomized, double-blind study between experimental prophylactic treatment with Lycopene vs placebo:

* Treatment A - lycopene tablets 20 mg
* Treatment B - placebo tablets

Patients should take orally Lycopene/placebo after dinner (to promote its absorption), starting the day before the beginning of treatment with panitumumab for the entire duration of the therapy, until progression of the disease or definitive drug suspension for toxicity.

Objectives of the study

Primary objective: to assess the effectiveness of lycopene versus placebo in reducing skin toxicity induced by panitumumab in patients treated for metastatic colorectal carcinoma.

Secondary objective: to assess lycopene pharmacokinetics

Exploratory objectives: to assess lycopene effectiveness versus placebo in increasing panitumumab effectiveness in terms of Disease Control (DC), Objective Response (OR) and Stabilisation of the Disease (SD). To assess lycopene effectiveness versus placebo in increasing panitumumab effectiveness in terms of Progression Free Survival (PFS).

As far as randomization is concerned, the two groups will be balanced according to sex, therapeutic line and institution in which patients will be treated.

ELIGIBILITY:
Standard schedules of these treatments would be used.

Inclusion and exclusion criteria would be the following:

Inclusion criteria:

1. Age ≥ 18 years;
2. Patients suffering from colorectal adenocarcinoma at stage-IV, for which a treatment with panitumumab is required;
3. No previous treatment with anti-EGFR drugs;
4. Presence of at least one neoplastic lesion one-dimensionally measurable;
5. No systemic anti-neoplastic therapy, nor experimental therapy or radiotherapy during the three weeks before randomization;
6. Proper contraceptive treatment by patient and his/her partner;
7. Written informed consent for participating to the study;
8. Performance Status (under ECOG scale) 0, 1. 2.

Exclusion criteria

1. PS > 2
2. Poor patient compliance;
3. Dermatological ongoing pathologies which contraindicate the treatment or made skin toxicity assessment difficult;
4. Presence of clinical conditions which could alter lycopene absorption (altered intestinal transit, malabsorption);
5. Pregnancy;
6. Absence of measurable lesions;
7. Previous treatment with anti-EGFR drugs;
8. Intolerance/allergy to tomato or milk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-08-03 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Skin toxicity reduction | Skin toxicity will be verified every two weeks assessed up to 12 weeks, from date of randomization until the date of first documented progression
  Reduction of grade 2/4 skin toxicity of 30% in the experimental group.
  Toxicity will be evaluated as:
  1. worst toxicity for each patient during the treatment;
  2. grade 3 or grade 4 toxicity duration related to the treatment duration for each patient in the two arms;
  3. number and duration of tetracyclines and antibiotic treatment related to the treatment duration for each patient in the two arms;
  4. toxicity in difference time points (G15, G29, .....) for each clinical skin features (rash papular, pustular - xerosis skin - paronychia) in the two arms

CONTACTS AND LOCATIONS:
Locations (1):
- Marco Pirovano, Milan, Italy

REFERENCES:
- [Result] Hu JC, Sadeghi P, Pinter-Brown LC, Yashar S, Chiu MW. Cutaneous side effects of epidermal growth factor receptor inhibitors: clinical presentation, pathogenesis, and management. J Am Acad Dermatol. 2007 Feb;56(2):317-26. doi: 10.1016/j.jaad.2006.09.005. Epub 2006 Dec 1. PMID 17141360
- [Result] Galimont-Collen AF, Vos LE, Lavrijsen AP, Ouwerkerk J, Gelderblom H. Classification and management of skin, hair, nail and mucosal side-effects of epidermal growth factor receptor (EGFR) inhibitors. Eur J Cancer. 2007 Mar;43(5):845-51. doi: 10.1016/j.ejca.2006.11.016. Epub 2007 Feb 7. PMID 17289377
- [Result] Pastore S, Mascia F, Mariani V, Girolomoni G. The epidermal growth factor receptor system in skin repair and inflammation. J Invest Dermatol. 2008 Jun;128(6):1365-74. doi: 10.1038/sj.jid.5701184. Epub 2007 Nov 29. PMID 18049451
- [Result] Rodeck U. Skin toxicity caused by EGFR antagonists-an autoinflammatory condition triggered by deregulated IL-1 signaling? J Cell Physiol. 2009 Jan;218(1):32-4. doi: 10.1002/jcp.21585. PMID 18781585
- [Result] Requena C, Llombart B, Sanmartin O. Acneiform eruptions induced by epidermal growth factor receptor inhibitors: treatment with oral isotretinoin. Cutis. 2012 Aug;90(2):77-80. PMID 22988651
- [Result] Chen J, Song Y, Zhang L. Effect of lycopene supplementation on oxidative stress: an exploratory systematic review and meta-analysis of randomized controlled trials. J Med Food. 2013 May;16(5):361-74. doi: 10.1089/jmf.2012.2682. Epub 2013 Apr 30. PMID 23631493
- [Result] Misale S, Di Nicolantonio F, Sartore-Bianchi A, Siena S, Bardelli A. Resistance to anti-EGFR therapy in colorectal cancer: from heterogeneity to convergent evolution. Cancer Discov. 2014 Nov;4(11):1269-80. doi: 10.1158/2159-8290.CD-14-0462. Epub 2014 Oct 7. PMID 25293556
- [Result] Lemieux E, Cagnol S, Beaudry K, Carrier J, Rivard N. Oncogenic KRAS signalling promotes the Wnt/beta-catenin pathway through LRP6 in colorectal cancer. Oncogene. 2015 Sep 17;34(38):4914-27. doi: 10.1038/onc.2014.416. Epub 2014 Dec 15. PMID 25500543
- [Result] Kim M, Jho EH. Cross-talk between Wnt/beta-catenin and Hippo signaling pathways: a brief review. BMB Rep. 2014 Oct;47(10):540-5. doi: 10.5483/bmbrep.2014.47.10.177. PMID 25154721
- [Result] Kahn M. Can we safely target the WNT pathway? Nat Rev Drug Discov. 2014 Jul;13(7):513-32. doi: 10.1038/nrd4233. PMID 24981364
- [Result] Khuda-Bukhsh AR, Das S, Saha SK. Molecular approaches toward targeted cancer prevention with some food plants and their products: inflammatory and other signal pathways. Nutr Cancer. 2014;66(2):194-205. doi: 10.1080/01635581.2014.864420. Epub 2013 Dec 30. PMID 24377653
- [Result] Stahl W, Sies H. beta-Carotene and other carotenoids in protection from sunlight. Am J Clin Nutr. 2012 Nov;96(5):1179S-84S. doi: 10.3945/ajcn.112.034819. Epub 2012 Oct 10. PMID 23053552
- [Result] Di Franco R, Calvanese M, Murino P, Manzo R, Guida C, Di Gennaro D, Anania C, Ravo V. Skin toxicity from external beam radiation therapy in breast cancer patients: protective effects of Resveratrol, Lycopene, Vitamin C and anthocianin (Ixor(R)). Radiat Oncol. 2012 Jan 30;7:12. doi: 10.1186/1748-717X-7-12. PMID 22289566
- [Result] Kasdagly M, Radhakrishnan S, Reddivari L, Veeramachaneni DN, Vanamala J. Colon carcinogenesis: influence of Western diet-induced obesity and targeting stem cells using dietary bioactive compounds. Nutrition. 2014 Nov-Dec;30(11-12):1242-56. doi: 10.1016/j.nut.2014.02.016. Epub 2014 Mar 12. PMID 25280404
- [Result] Li Y, Wicha MS, Schwartz SJ, Sun D. Implications of cancer stem cell theory for cancer chemoprevention by natural dietary compounds. J Nutr Biochem. 2011 Sep;22(9):799-806. doi: 10.1016/j.jnutbio.2010.11.001. Epub 2011 Feb 4. PMID 21295962
- [Result] Preet R, Mohapatra P, Das D, Satapathy SR, Choudhuri T, Wyatt MD, Kundu CN. Lycopene synergistically enhances quinacrine action to inhibit Wnt-TCF signaling in breast cancer cells through APC. Carcinogenesis. 2013 Feb;34(2):277-86. doi: 10.1093/carcin/bgs351. Epub 2012 Nov 5. PMID 23129580
- [Result] Sarkar FH, Li Y, Wang Z, Kong D. The role of nutraceuticals in the regulation of Wnt and Hedgehog signaling in cancer. Cancer Metastasis Rev. 2010 Sep;29(3):383-94. doi: 10.1007/s10555-010-9233-4. PMID 20711635
- [Result] Tang FY, Pai MH, Wang XD. Consumption of lycopene inhibits the growth and progression of colon cancer in a mouse xenograft model. J Agric Food Chem. 2011 Aug 24;59(16):9011-21. doi: 10.1021/jf2017644. Epub 2011 Jul 25. PMID 21744871
- [Result] Tang FY, Shih CJ, Cheng LH, Ho HJ, Chen HJ. Lycopene inhibits growth of human colon cancer cells via suppression of the Akt signaling pathway. Mol Nutr Food Res. 2008 Jun;52(6):646-54. doi: 10.1002/mnfr.200700272. PMID 18537129
- [Result] Shao A, Hathcock JN. Risk assessment for the carotenoids lutein and lycopene. Regul Toxicol Pharmacol. 2006 Aug;45(3):289-98. doi: 10.1016/j.yrtph.2006.05.007. Epub 2006 Jun 30. PMID 16814439
- [Result] Lacouture ME, Maitland ML, Segaert S, Setser A, Baran R, Fox LP, Epstein JB, Barasch A, Einhorn L, Wagner L, West DP, Rapoport BL, Kris MG, Basch E, Eaby B, Kurtin S, Olsen EA, Chen A, Dancey JE, Trotti A. A proposed EGFR inhibitor dermatologic adverse event-specific grading scale from the MASCC skin toxicity study group. Support Care Cancer. 2010 Apr;18(4):509-22. doi: 10.1007/s00520-009-0744-x. Epub 2010 Feb 10. PMID 20145956
- [Result] Douillard JY, Siena S, Cassidy J, Tabernero J, Burkes R, Barugel M, Humblet Y, Bodoky G, Cunningham D, Jassem J, Rivera F, Kocakova I, Ruff P, Blasinska-Morawiec M, Smakal M, Canon JL, Rother M, Oliner KS, Tian Y, Xu F, Sidhu R. Final results from PRIME: randomized phase III study of panitumumab with FOLFOX4 for first-line treatment of metastatic colorectal cancer. Ann Oncol. 2014 Jul;25(7):1346-1355. doi: 10.1093/annonc/mdu141. Epub 2014 Apr 8. PMID 24718886